CLINICAL TRIAL: NCT04763889
Title: Feasibility Study of a Short Term Cognitive Behaviour Therapy Intervention Targeting Anxiety and Coping Styles for Adults With Allergy.
Brief Title: Cognitive Behaviour Therapy for Adults With Allergy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHMS 20-21 006 EGA
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-08

CONDITIONS: Allergy; Anxiety
MeSH Terms: conditions — Hypersensitivity; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT workshop (Experimental): Participants will be randomly allocated to either a self-help control group or a CBT workshop group. In the intervention group participants will attend a day workshop or two half day workshops focused on using CBT to manage their anxiety and stress.
  Interventions: Behavioral: CBT
- Self-help control treatment as usual group (No Intervention): Participants will be randomly allocated to either a self-help control group or a CBT workshop group. Participants in the treatment as usual group will receive the workshop materials after the active treatment group have completed their final follow-up at 3 months

INTERVENTIONS:
Behavioral: CBT — CBT for those with an allergy and anxiety
  Arms: CBT workshop

SUMMARY:
People with severe allergy often experience distress but research exploring psychological interventions for them is limited. Cognitive Behaviour Therapy (CBT) is routinely used in NHS services. The research investigators would like to know whether a short term CBT group is feasible and acceptable for those with severe allergy who are also experiencing distress and/or anxiety.

The research investigators will recruit people with allergy through support groups and social media. Those interested in the study will be invited to complete a screening interview. If the participants meet the inclusion criteria and consent to take part the participants will be randomly allocated into the CBT or a self-help group. Full written consent will be needed at the telephone screening session if participants are eligible for the study. Participants will be given time to complete this prior to the intervention. Participants will be able to withdraw at any point during the study.

The self-help group will be sent self-help materials. The CBT group will attend a single session day workshop based on CBT (maximum 6 hours length). Due to the Covid-19 pandemic, the workshop may need to be delivered online. If delivered online, the workshop may be delivered over two three hour sessions.

Participants will be asked to complete questionnaires at baseline, the day of the intervention, one month later and three months later. They will be asked to complete a feedback form about their experiences in the group and at three month follow up, a small subsample of participants will be invited to interview.

Once the data is analysed it will be written up into a report for a clinical psychology doctoral qualification major research project. It may also be published in academic journals and presented at conferences. A possible outcome of the research is that people with allergy either do or do not find the workshops an acceptable and/or feasible intervention. It will identify the potential for this intervention to reduce distress and anxiety and to improve coping skills in adults with allergy. Those who take part are welcome to contact the researchers to find out the results of the study.

DETAILED DESCRIPTION:
Background Adults with severe allergy often experience distress but research exploring psychological interventions for this group has not been carried out. Cognitive Behaviour Therapy has previously been found to reduce distress in mothers of children with severe allergy. Indeed, there are two allergy specialist clinics in the UK which offer interventions to children and families with severe allergy. Initial investigations have shown these clinics to be beneficial. It is clear that a study is needed to explore the feasibility of a CBT intervention for adults with severe allergy in order for further research to be conducted and to improve outcomes for this group.

The feasibility study will involve recruiting adults with severe allergy and inviting them to screening interview phone call. If suitable for the study, participants will be randomly allocated to an intervention or control group. Those in the intervention group will be invited to attend a single session 6 hour workshop focusing on adapted CBT for allergy. There is evidence that single session workshops can be beneficial in managing anxiety. The workshop in the current study will either be face to face groups or due to the Covid-19 pandemic, the workshops may be delivered on online platforms, such as Zoom. If delivered online, the workshop will likely to be split over two three hour sessions. Online delivery of the intervention may be more beneficial for those with disabilities, who may be at a higher risk of experiencing complications due to the Coronavirus i.e. those with allergy and asthma. Indeed, delivery online would lead to flexibility for participants who may be located across the UK without needing to travel long distances. Those who have long term health problems may prefer the flexibility of online delivery as this limits their need to travel. This may also suit parents who would not necessarily need childcare arrangements for an online workshop.

Those in the control group will be sent self-help information. Questionnaire measures will explore quality of life, coping style, anxiety, worry, stress and depression. Questionnaires will also explore personal goals for therapy and self-care behaviours. With questionnaire measures, reliable change and the proportion meeting 'clinical caseness' pre and post intervention will be explored to provide a signal of efficacy of the intervention. Changes between the groups will also be assessed. As the study is assessing feasibility, retention and uptake will be assessed. Feedback questionnaires at the end of the study, including free text responses and Likert Scale questionnaires, will also be collected to assess acceptability and to explore participant experiences of the study. Additionally, qualitative interviews with a small subsample of participants being followed up after three months will also be conducted to assess acceptability. The interviews will focus on participants experiences of living with an allergy and the experience of the workshop and research.

Aims of the study

The study's objective is to assess the feasibility and acceptability of a short term CBT group intervention for reducing anxiety and distress in those with severe allergy. The research questions are:

* Can appropriate participants be recruited and retained to the group intervention?
* How appropriate are the data collection procedures and outcome measures for the participants and purposes of the study?
* Are study procedures and workshop intervention suitable for and acceptable to participants?
* What is it like to attend a group intervention for people with severe allergy and anxiety/distress?
* Does the intervention provide a signal of efficacy to warrant a definitive trial?

Method Participants with allergy will be recruited through support groups and social media. Those who are interested in the study will be asked to complete a screening interview. If they meet inclusion criteria and consent to take part they will be randomly allocated into either an intervention or a control group. The intervention group will attend a single session day workshop based on CBT. The control group will be sent self-help materials. Due to the Covid-19 pandemic, the workshop may need to be delivered online. If delivered online, the workshop may be delivered over two sessions. Participants will be asked to complete feedback forms about their experiences in the group. At three month follow up, a small subsample of participants will be interviewed. The interviews will focus on participants experiences of living with an allergy and the experience of the workshop and research.

Results A possible outcome is that people with allergy and emotional distress either do or do not find the workshops an acceptable and feasible intervention. It will identify dropout rates and participant retention. It will also identify the potential for this intervention to reduce distress and anxiety and to improve coping skills in adults with severe allergy.

Implications If the outcome of the study is that CBT is an acceptable intervention for those with severe allergy and emotional distress, it adds weight to the argument that more research is needed to explore this on a larger scale. If the outcome measures are acceptable for this client group, they could be used in a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 upwards.
* Adults with an allergy diagnosed both as adults and as children.
* Adults with an allergy who report experiencing emotional distress.
* Participant is able to attend a day workshop session (6 hours maximum). This will either be delivered face to face or due to the Covid-19 pandemic these may need to be delivered online (i.e. via Zoom) rather than face to face. If this is the case the workshop may be split into two three hourly sessions. Therefore, the participant would need access to a computer, smart phone or tablet and have access to the internet.

Exclusion Criteria:

* Participant does not speak English.
* Participant is unable to have the capacity to provide informed consent.
* Participant is taking part in another interventional study.
* Those with severe psychological difficulties and co-morbidities, such as active psychosis, a diagnosis of a personality disorder, schizophrenia and bipolar disorder or is receiving care from mental health team.
* Those who may not be able to engage cognitively with the workshop materials and questionnaires (i.e. those with a significant learning disability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Change in the Food Allergy Quality of Life Questionnaire- Adult Form (FAQLQ-AF, Flokstra-de Blok et al., 2009) | Questionnaires will be given at baseline, 1 month and at 3 month follow up.
  Questionnaire

SECONDARY OUTCOMES:
Change in Penn State Worry Questionnaire (PSWQ, Meyer et al., 1990) | Questionnaires will be given at baseline, 1 month and at 3 month follow up.
  Questionnaire
Change in Depression, Anxiety and Stress Scale-21 (DASS 21, Lovibond & Lovibond, 1995) | Questionnaires will be given at baseline, 1 month and at 3 month follow up.
  Questionnaire. 21 items. Rate on a scale from 0-3 how much each statement applied to them. Three factors: depression, anxiety and stress. The higher the score the higher the levels of depression, anxiety and stress.
Change in the COPE scale (Carver, Scheier & Weintraub, 1989) | Questionnaires will be given at baseline, 1 month and at 3 month follow up.
  Questionnaire. 60 items. Participants rate on a 4 point Likert Scale (1-4). This measures 15 coping strategies and 4 factors including problem focused, emotion focused, avoidance focused and acceptance focused coping. There is no 'overall score' for this measure but higher scores on specific coping styles suggesting more use of this.
Change in Self-care Likert Scale (Jones et al., 2014) | Questionnaires will be given at baseline, 1 month and at 3 month follow up.
  Questionnaire. Five items. Responses are measured on a 6-point scale (0-5) how much each statement applies to them. Higher the score suggests poorer self-care behaviours.
Change in Goal based outcome measure: clients will be asked to choose a goal at the start of the workshop and rate how well they have achieved that by the end on a 0-10 scale (0 = worst, 10 = best) | Questionnaires will be given immediately post-intervention, after 1 month and at 3 month follow up.
  Questionnaire

OTHER OUTCOMES:
Interview | At three month follow up
  Semi-structured interview
Demographic information | Collected at baseline
  Demographic questionnaire
Feedback survey | At 3 month follow up
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jones, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung MC, Walsh A, Dennis I. Trauma exposure characteristics, past traumatic life events, coping strategies, posttraumatic stress disorder, and psychiatric comorbidity among people with anaphylactic shock experience. Compr Psychiatry. 2011 Jul-Aug;52(4):394-404. doi: 10.1016/j.comppsych.2010.09.005. Epub 2010 Nov 16. PMID 21081226
- [Background] Knibb RC. Effectiveness of Cognitive Behaviour Therapy for Mothers of Children with Food Allergy: A Case Series. Healthcare (Basel). 2015 Nov 25;3(4):1194-211. doi: 10.3390/healthcare3041194. PMID 27417820
- [Background] Knibb R, Halsey M, James P, du Toit G, Young J. Psychological services for food allergy: The unmet need for patients and families in the United Kingdom. Clin Exp Allergy. 2019 Nov;49(11):1390-1394. doi: 10.1111/cea.13488. Epub 2019 Sep 8. PMID 31454459
- [Background] Cartwright-Hatton S, Ewing D, Dash S, Hughes Z, Thompson EJ, Hazell CM, Field AP, Startup H. Preventing family transmission of anxiety: Feasibility RCT of a brief intervention for parents. Br J Clin Psychol. 2018 Sep;57(3):351-366. doi: 10.1111/bjc.12177. Epub 2018 Mar 25. PMID 29575043
- [Background] Flokstra-de Blok BM, van der Meulen GN, DunnGalvin A, Vlieg-Boerstra BJ, Oude Elberink JN, Duiverman EJ, Hourihane JO, Dubois AE. Development and validation of the Food Allergy Quality of Life Questionnaire - Adult Form. Allergy. 2009 Aug;64(8):1209-17. doi: 10.1111/j.1398-9995.2009.01968.x. Epub 2009 Feb 11. PMID 19210345
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Jones CJ, Smith HE, Frew AJ, Toit GD, Mukhopadhyay S, Llewellyn CD. Explaining adherence to self-care behaviours amongst adolescents with food allergy: a comparison of the health belief model and the common sense self-regulation model. Br J Health Psychol. 2014 Feb;19(1):65-82. doi: 10.1111/bjhp.12033. Epub 2013 Feb 12. PMID 23398539
- [Derived] Jones CJ, Tallentire H, Edgecumbe R, Sherlock G, Hale L. Online, group, low-intensity psychological intervention for adults, children, and parents with food allergy. Ann Allergy Asthma Immunol. 2024 Oct;133(4):453-461. doi: 10.1016/j.anai.2024.07.025. Epub 2024 Jul 26. PMID 39069154
- See also: Lovibond, S. H., & Lovibond, P. F. (1995). Manual for the depression anxiety stress scales (2nd ed.). Sydney: Psychology Foundation. — http://www2.psy.unsw.edu.au/dass/order.htm